CLINICAL TRIAL: NCT06406361
Title: The Effect of an Online Stres Management Program on the Individual Workload Perception and Stress of Nurses: A Non-randomized Quasi-experimental Design Study
Brief Title: The Effect of Online Stress Management Program on Nurses' Individual Workload Perception, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Gozde Yıldız Daş Geçim, Assist. Prof., Amasya University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AmasyaU28
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stress Management; Stress; Nursing
Keywords: stress management program; individual workload perception; stress; nursing

STUDY DESIGN:
Intervention Model Description: a pretest-posttest control group design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A total of six-sessions of Online Stress Management program were applied to the experimental group, consisting of 40-50 minutes and one sessions per week.
  Interventions: Behavioral: online stress management program
- control group (No Intervention): not intervention

INTERVENTIONS:
Behavioral: online stress management program — -Nurses should have an idea about stress management program Awareness develops about the importance of attending sessions regularly. Nurses have information about the training program. Joint session dates are determined. The educator makes statements about himself and education. The benefits of education for nurses are explained. Nurses are informed about the general rules of education. The importance of regular attendance at sessions is emphasized. Privacy rules and limits are determined. The necessity of completing homework is explained. Nurses are enabled to share their feelings and thoughts. Ensuring that nurses are able to recognize stress and reactions to stress and identify sources of stress in individual and business life.
  Being informed about the effects of stress and negative workload perception Being able to recognize the tension created by stress in the body Learning breathing and deep relaxation techniques to reduce or eliminate symptoms of stress
  Arms: Experimental group

SUMMARY:
Negative workload perception and stress are very important issues in occupational health. The aim of this study is to evaluate the effect of Online Stress Management (OSM) program on nurses' individual workload perception, and stress. The study included 90 nurses who met the inclusion criteria and signed the informed consent form. In the study, 45 nurses were allocated to the experimental group and 45 nurses were allocated to the control group. Due to the intensive working conditions of the nurses, staff shortages, workload, and restrictions such as shift work, participants could not be randomly assigned to the groups. Nurses who agreed to participate in the OSM program were voluntarily assigned to the experimental group, and those who did not want to participate were assigned to the control group.

DETAILED DESCRIPTION:
Introduction: The feeling of stress and individual workload perception are an uncomfortable situation for individuals, are important factors that affect the physical and mental health and quality of life of health professional. Perception of workload and stress, which are basic elements in the field of occupational health, are important factors in coping with problems arising from working conditions and increasing the efficiency of work. Increased individual workload perception and stress are quite common, especially in nurses with intense working conditions.

Aim: The aim of the study was to investigate the effect of stress management training on nurses' individual workload perception and stress using a non-randomized, waiting list comparison design.

Methods: The analyses included a total of 86 nurses (experimental group n = 42 and control group n = 44). A total of six-sessions of OSM program were applied to the experimental group, consisting of 40-50 minutes and one sessions per week. Data were collected using the 'Participant Information Form', 'Nurse Stress Scale' (NSS) and 'Individual Workload Perception Scale' (IWPS). Time and group changes in stress, and individual workload perception were computed using a repeated measures analysis of variance (ANOVA) model was used to test the between-group differences from baseline to six weeks.

ELIGIBILITY:
Inclusion Criteria:

* being a nurse
* were working in the institution at the time of the study;
* not have visual or hearing disorders;
* not have any diagnosed chronic disease that potentially
* prevented participation in the study; did not have a mental health problem;
* agreed to participate in the study.

Exclusion Criteria:

* have a known physical or neurological disease
* not working in the institution at the time of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Nurse Stress Scale | at the end of the 1 months
  The NSS total scores range from 34-136. The total score measures the frequency of stress experienced by a nurse and can be calculated by adding the participant's responses to all items. The high overall score indicates that the nurse experiences more frequent stress periods about individual stress problems in the physical, psychological, and physical environment. A lower score indicates that the nurse experiences less stress for the same situations

SECONDARY OUTCOMES:
Individual Workload Perception Scale | at the end of the 1 months
  The lowest total score that can be obtained from the scale is 31 and the highest is 155. As the score obtained from the scale increases, the individual workload perception is evaluated positively.

CONTACTS AND LOCATIONS:
Overall Officials: nihan yalciner durgu, PhD, Study Chair — Manisa Celâl Bayar University
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No